CLINICAL TRIAL: NCT03909074
Title: A Phase III Clinical Trial With Randomized, Double-blinded, Controlled Design as Well as Bridging Design to Evaluate the Safety and Immunogenicity of EV71 Vaccine in Children Aged 36-71 Months
Brief Title: Clinical Trial of Enterovirus 71（EV71） Inactivated Vaccine in Children Aged 36-71 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-EV71-3003
Record Dates: First submitted 2019-03-29; First posted 2019-04-09 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2020-01

CONDITIONS: Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): 36-71 months old children-experimental EV71 vaccine.
  Interventions: Biological: 36-71 months old children-experimental EV71 vaccine.
- Vaccine-controlled group (Active Comparator): 36-71 months old children-control EV71 vaccine.
  Interventions: Biological: 36-71 months old children-control EV71 vaccine.
- Age-controlled group (Active Comparator): 6-35 months old children-experimental EV71 vaccine.
  Interventions: Biological: 6-35 months old children-experimental EV71 vaccine.

INTERVENTIONS:
Biological: 36-71 months old children-experimental EV71 vaccine. — Two doses experimental EV71 vaccine at the 0, 30 days vaccination schedule.
  Arms: Experimental group
Biological: 36-71 months old children-control EV71 vaccine. — Two doses control EV71 vaccine at the 0, 30 days vaccination schedule.
  Arms: Vaccine-controlled group
Biological: 6-35 months old children-experimental EV71 vaccine. — Two doses experimental EV71 vaccine at the 0, 30 days vaccination schedule.
  Arms: Age-controlled group

SUMMARY:
The purpose of this study is to evaluate the non-inferiority of experimental EV71 vaccine compared to the control EV71 vaccine in children aged 36-71 months, to evaluate the non-inferiority of EV71 vaccine used in children aged 36-71 months compared to 6-35 months. The experimental vaccine was manufactured by Sinovac Biotech Co., Ltd, and the control vaccine was manufactured by Institute of Medical Biology Chinese Academy of Medical Sciences.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, single-center, controlled phase III clinical trial in children aged 36-71 months, and bridging trial between agegroup of 6-35 and 36-71 months. The purpose of this study is to evaluate the immunogenicity and safety of the experimental EV71 vaccine in children aged 36-71 months. The primary objective of this study is to evaluate the non-inferiority of experimental EV71 vaccine compared to the control EV71 vaccine in children aged 36-71 months, and the non-inferiority of EV71 vaccine used in children aged 36-71 months compared to 6-35 months. The secondary objective is to evaluate the safety of the experimental vaccine used in children aged 36-71 months. The experimental vaccine is manufactured by Sinovac Biotech Co., Ltd, and the control vaccine is manufactured by Institute of Medical Biology Chinese Academy of Medical Sciences. 600 children aged 36-71 months will be randomly assigned in to receive the experimental vaccine or control vaccine, and 300 children aged 6-35 months will receive the experimental vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ≥ 2 years old;
* Proven legal identity;
* Participants or guardians of the participants should be capable of understanding the written consent form, and such form should be signed prior to enrolment.

Exclusion Criteria:

* Prior vaccination with EV71 vaccine;
* History of hand, foot and mouth disease;
* History of allergy to any vaccine or vaccine ingredient, asthma, serious adverse reactions to vaccination, such as urticaria, dyspnea, angioneurotic edema, abdominal pain, etc;
* Congenital malformation, developmental disorders, genetic defects, or severe malnutrition;
* Autoimmune disease or immunodeficiency/immunosuppressive;
* Severe/uncontrollable nervous system disease (epilepsy, seizures or convulsions) or mental illness;
* History of thyroidectomy, no spleen and functional spleen;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders;
* Receipt of any of the following products:

  1. Any immunosuppressant, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) within 6 month prior to study entry
  2. Blood products within 2 months prior to study entry
  3. Any other investigational products (drug or vaccine）within 30 days prior to study entry
  4. Any live attenuated vaccine within 14 days prior to study entry
  5. Any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Axillary temperature > 37.0 °C;
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
The seroconversion rates (SCR) of the EV71 neutralizing antibody calculated based on the cutoff value of 1:8 | 30 days after two doses
  Subjects whose pre-immune antibody titer < 1:8 and post-immune antibody titer ≥ 1:8, or those whose pre-immune antibody titer ≥ 1:8 and the increase of post-immune antibody level ≥ 4 folds are considered seroconverted.
The Geometric mean titer (GMT) of the EV71 neutralizing antibody in the susceptible population | 30 days after two doses
  The susceptible population refer to the subjects whose pre-immune antibody titer <1:8

SECONDARY OUTCOMES:
The overall incidence of adverse reactions | 0-30 days after each dose
  After each dose, a 30-minute safety observation will be conducted immediately. The body temperature, solicited local and general adverse events (AE) on day 0-7 were reported. The solicited local symptoms include pain, induration, redness, swelling, rash, and pruritus. The solicited general adverse symptoms include allergy, fatigue, irritability, inappetence, vomiting, diarrhea, and fever. Unsolicited adverse events on day 0-30 were also reported, which include the unsolicited symptoms happened within 0-7 days, and any symptoms happened within the 8-28 days. Each AE case will be reviewed by the investigator to determine whether it was an adverse reaction (The vaccination-related AE). The incidence of adverse reactions=Number of subjects who have adverse reactions of any symptoms/number of all the subjects whose safety information are collected.
The incidence of the serious adverse events (SAE) | 0-30 days after each dose
  After each dose, the serious adverse events in the safety observation period will be reported. The SAE incidence=Number of subjects who have SAE of any symptoms/Number of subjects whose safety information are collected.
The seroconversion rates (SCR) of the EV71 neutralizing antibody calculated based on the cutoff value of 1:16, 1:32, and 1:64 respectively | 30 days after two doses
  Subjects whose pre-immune antibody titer <1:16(1:32/1:64) and post-immune antibody titer ≥1:16(1:32/1:64), or those whose pre-immune antibody titer ≥ 1:16(1:32/1:64) and the increase of post-immune antibody level ≥ 4 folds are considered seroconverted.
The Geometric mean titer (GMT) of the EV71 neutralizing antibody | 30 days after two doses
  The GMT 30 days after two doses.

CONTACTS AND LOCATIONS:
Overall Officials: Lifen Zhang, Master, Principal Investigator — Yunnan Center for Disease Control and Prevention
Locations (1):
- Yun County Center for Disease Control and Prevention, Lincang, Yunnan, China

REFERENCES:
- [Derived] Zhang L, Gao F, Zeng G, Yang H, Zhu T, Yang S, Meng X, Mao Q, Liu X. Immunogenicity and Safety of Inactivated Enterovirus 71 Vaccine in Children Aged 36-71 Months: A Double-Blind, Randomized, Controlled, Non-inferiority Phase III Trial. J Pediatric Infect Dis Soc. 2021 Apr 30;10(4):440-447. doi: 10.1093/jpids/piaa129. PMID 33269798